CLINICAL TRIAL: NCT02868151
Title: Effect of Ascorbic Acid Oral Supplementation in Assessing the Severity of Oral Mucositis in Chemo-radiation Therapy of Head and Neck Cancers.
Brief Title: Effect of Oral Vitamin C in Assessing the Severity of Oral Mucositis in Chemoradiation of Head and Neck Cancers
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre (Other)
Collaborators: Saveetha University (Other); MNJ Institute of Oncology and Regional Cancer Center (Other Government)
Responsible Party: Principal Investigator, NALLAN CHAITANYA, Associate Professor, department of oral medicine and radiology, panineeya institute of dental sciences, Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ECR/227/INSP/AP/2014
Record Dates: First submitted 2016-08-06; First posted 2016-08-16 (Estimated); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Oral Mucositis
Keywords: Oral mucositis, chemo radiotherapy, vitamin c,
MeSH Terms: conditions — Stomatitis | interventions — Ascorbic Acid; Zinc Acetate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- GROUP A (No Intervention): Standard treatment followed in the regional cancer center for prevention and treatment of oral mucositis during chemo radiotherapy of cancers. 20% Benzocaine 15grms. twice daily for the entire treatment period
- GROUP B (Experimental): Ascorbic acid oral supplementation 1g four times daily for the entire treatment period of 30 days and after treatment by tapering the dose of the drug to half for another month. The drug has to be started 2 days prior to initiation of treatment of cancer.
  Subdivided into 2 groups , 30 patients in each : sub group 1: only radiotherapy patients, subgroup 2 includes concurrent chemo-radiotherapy patients.
  Interventions: Drug: Ascorbic Acid
- GROUP C (Experimental): Zinc acetate tablets 50mg orally
  Interventions: Drug: Zinc acetate

INTERVENTIONS:
Drug: Ascorbic Acid — Ascorbic acid oral supplementation 1g four times daily for the entire treatment period and 30 days after treatment by tapering the dose of the drug to half. The drug has to be started 2 days prior to initiation of treatment of cancer.
  Other Names: Vitamin C
  Arms: GROUP B
Drug: Zinc acetate — Zinc acetate 50mg tablets orally twice daily for entire period of cancer treatment
  Arms: GROUP C

SUMMARY:
The surrounding controversies both advocating and simultaneously opposing the use of vitamin C, mostly extrapolating animal models to human models, it has not been used individually to assess the severity of oral mucositis during chemoradiotherapy.

The present study is undertaken to evaluate the effect of vitamin C oral supplements in assessing the severity of oral mucositis during chemoradiotherapy for oral cancer.

DETAILED DESCRIPTION:
Oral mucositis is a predictable and unavoidable representation during the course of radiotherapy employed for treatment of head and neck cancers. The term oral mucositis is used to describe inflammation of the oral mucosa, a separate entity distinct from oral lesions with other pathogenic background generally summarized as stomatitis. The cells that line the gastrointestinal tract from the mouth to the rectum are especially vulnerable to such changes. The incidence and severity of oral mucositis is influenced by the type of antineoplastic treatment administered and patient related factors. The pathogenesis of radiation mucositis though not completely understood, is usually either by direct DNA damage or via an indirect mechanism of releasing free radicals upon radiolysis of water effecting the oral epithelium.It is associated with significant morbidity, pain, odynophagia, malnutrition thereby affecting the overall quality of life in these patients and carrying a more important risk of systemic infections particularly in impaired host defense setup.In addition to acute damage wide range of GI mucosal involvement occurs during radiotherapy.

Various radiation modifying agents have been used which can either selectively protect normal cells but not tumor cells against therapeutic damage or can selectively enhance the effect of radiation on tumor cells but not on normal cells thereby improving efficacy of radiation therapy. In spite of extensive research most of them are found to be toxic.

Antioxidants represent most selective radiation modifying agents that are non toxic to humans. However, because of many conflicting hypothesis on their usage affecting tumor response and also decreasing the radiation induced toxicity on normal cells, recommendations have followed for their non usage during chemo-radiotherapy. In spite of such reservations on behalf of oncologists over 70% of patients are on antioxidant supplements such as those containing vitamin A, vitamin C and polar carotenoids with or without the knowledge of oncologists.

Antioxidants can neutralize those free radicals generated during radio-chemo therapy enhancing body's antioxidant stores in order to prevent mucositis and to maintain healthy oral tissues. Literature survey provides exhaustive list of such antioxidants successfully implicated in controlling oral mucositis to some extent. Antioxidants such as beta carotene, vitamin E and vitamin C in combination, glutamine, glutathione have been studied.

Vitamin C is a water soluble nutrient that has wide antioxidant and wound healing properties. It has been widely in scurvy patients but its effect on conventional cancer therapy by radiation and chemotherapy were little known. Limited preclinical data suggested that this vitamin at high concentrations increased the toxicity of certain chemotherapeutic drugs in animals.

Recommended daily allowance (RDA) for vitamin C is 90mgper day for men and 75mg per day for women, upper limit being 2000mg per day. Evidence points out that the intake to achieve therapeutic tissue concentration in normal people should be several times higher than RDA. Conversely a recent study implicated dangers of consuming high doses of vitamin C which may turn from antioxidant to pro oxidant interfering radiotherapy. However it should be noted that the conditions used in the above study prevailed were invitro in nature, which cannot reflect an identical situation invivo. Few other studies believed that it can enhance immune function by increasing natural killer cells and lymphocyte activity.

With such controversial background and paucity of data in human intervention, this study is undertaken to evaluate the effect of vitamin c in assessing the severity of oral mucositis in patients undergoing cancer chemo and radiotherapy concurrently

ELIGIBILITY:
Inclusion Criteria:

All patients who are attending Mehdi Nawaz Jung cancer hospital for radiotherapy and who provide written consent for the study.

Exclusion Criteria:

* Patients with known allergy to vitamin C
* Patients with Glucose-6-phosphate dehydrogenase deficiency
* Patients with renal failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2016-08; Primary Completion 2017-12 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
World Health Organization criteria of grading oral mucositis.for head and neck cancer patients | one and half years.
  oral mucositis severity would be measured weekly in all the patients during the entire treatment of radiotherapy/chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: SANJEEVA KUMARI, MD, Principal Investigator — MNJ Institute of Oncology and Regional Cancer Center
Locations (1):
- MNJ institute of oncology & regional cancer center, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No
confidential data from hospital.